CLINICAL TRIAL: NCT02362386
Title: Feasibility of Obtaining Adipose Derived Regenerative Cells (ADRCs) From Discarded Thermal Burn Eschar Tissue Using Investigational Celution® System for Autologous Treatment of Thermal Burn Injury (The FAST Trial)
Brief Title: Feasibility of Obtaining ADRCs From Discarded Thermal Burn Eschar Tissue Using Investigational Celution® System
Status: Completed | Type: Observational
Sponsor: Cytori Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: The FAST Study
Record Dates: First submitted 2015-02-09; First posted 2015-02-12 (Estimated); Last update posted 2016-04-05 (Estimated); Status verified 2016-04

CONDITIONS: Thermal Burn

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Adipose tissue and adipose derived regenerative cells (ADRCs) will be obtained for microbiological testing and for non-DNA-based cell characterization.
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Celution Device — Non-interventional evaluation of Celution Device preparation of ADRCs from thermal burn eschar tissue that would normally be discarded.

SUMMARY:
The objective of the study is to assess the logistical and biological feasibility of preparing ADRCs from adipose tissue excised during standard-of-care burn wound excision using the Celution® System for autologous, same-day application to the burn wound.

DETAILED DESCRIPTION:
This study is a non-interventional clinical study. Adipose tissue excised as part of usual care of burn wound that would otherwise be discarded will be collected for processing and analysis. Target population includes patients with a burn injury that requires surgery in which fat excision of approximately 100 g (or more) is anticipated. The scope of the study includes:

* Fat tissue collected from tangential or fascial excision will be manually prepared for processing within the investigational Celution® System
* Adipose tissue will be processed using the investigational Celution® System. ADRC yield and viability will be evaluated using a NucleoCounter® device
* Age, gender, weight, height, location/severity/%TBSA of burn, time/date of burn injury, current stage of health will be collected
* Operational details such as start and stop time of tissue excision, adipose tissue preparation and Celution® processing, cell counting and dose preparation will be collected. In addition, weight of excised tissue prior to and after preparation, weight of adipose tissue processed by Celution Device and ADRC yield and viability will be recorded.
* Several samples will be collected and sent to a central microbiology laboratory for microbiological testing.

ELIGIBILITY:
Inclusion Criteria

1. Males or females ≤ 80 years of age
2. Admission to hospital for acute burn injury
3. Planned escharectomy anticipated to yield at least 100 g adipose tissue according to the treating surgeon's clinical judgment.

Exclusion Criteria

1. Known history of HIV infection, or has active Hepatitis B or active Hepatitis C infection
2. Pre-existing condition requiring current use of immunosuppressive medication or systemic steroids
3. Cancer requiring chemotherapy or radiation within previous 12 months

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Target population includes patients with a burn injury that requires surgery in which fat excision of approximately 100 g (or more) is anticipated
Sampling Method: Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2015-06; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Logistical Feasibility of Preparing ADRCs from discarded eschar tissue | 1 day
  Examine various parameters including time to assess how processing of adipose tissue using Celution Device could be integrated into standard-of-care thermal burn wound excision

SECONDARY OUTCOMES:
Cell Characterization | 1 day
  Cell viability, cell yield, non-DNA-based cell phenotype, microbiology

CONTACTS AND LOCATIONS:
Overall Officials: Steven Kesten, MD, Study Director — Cytori Therapeutics, Inc.
Locations (4):
- United States (4):
  - Arizona Burn Center at Maricopy Integrated Health Systems, Phoenix, Arizona
  - UC San Diego Medical Center, San Diego, California
  - University of Texas Medical Branch and Shriners Hospital for Children, Galveston, Texas
  - University ofWashington/Harborview Medical Center, Seattle, Washington